CLINICAL TRIAL: NCT05766397
Title: Evaluation of Occupational Exposure of Methoxyflurane to Paramedics in the Back of an Ontario, Canada Approved Ambulance.
Brief Title: Prehospital Inhaled Methoxyflurane Non-Clinical Occupational Exposure Study
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Mayday Fund (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CRRF 4869
Record Dates: First submitted 2023-02-21; First posted 2023-03-13 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Occupational Exposure
Keywords: paramedic; occupational exposure
MeSH Terms: interventions — Methoxyflurane

STUDY DESIGN:
Intervention Model Description: This is a phase other study. This is a phase other, Health Canada regulated, non-clinical occupational exposure laboratory study, where 30 healthy human participants will inhale methoxyflurane following a protocol and during which occupational exposure of methoxyflurane will be measured via strategically positioned samplers (active and passive) according to a pre-set protocol, including single and multiple consecutive events.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health volunteer (Other): Health volunteers will follow a standard protocol for inhalation of methoxyflurane while the off-gassing will be captured.
  Interventions: Drug: Methoxyflurane

INTERVENTIONS:
Drug: Methoxyflurane — Methoxyflurane belongs to the fluorinated hydrocarbon group of volatile anesthetic gases

SUMMARY:
Methoxyflurane is an anesthetic gas and at low doses has shown to help with pain. Methoxyflurane was approved in Canada in 2018. Low-dose methoxyflurane is self-administered by patients via a handheld inhaler. Exhaled methoxyflurane is captured by an activated carbon (AC) chamber fitted to the inhaler in order to minimize environmental and occupational exposure. It provides rapid (<1 minute), short-term (30-45 minutes) pain relief within six to ten inhalations and has been shown to be effective and safe in emergency care and for minor surgical, radiological, and dental procedures.

The current dosing recommendation is 3 ml bottle. However, the frequency at which methoxyflurane treatment can be safely used by paramedics is not established. From the product monograph, a patient's maximum daily dose of 6 mLs and weekly 15 mLs of methoxyflurane. The treatment course of methoxyflurane for patients should not be repeated at an interval of less than 3 months. Despite the activated carbon chamber to capture the exhaled methoxyflurane, when paramedics are supervising patients receiving inhaled analgesia within a confined area (like the back of an ambulance), it is possible that a paramedic may experience intermittent exposure to methoxyflurane vapour. Multiple use of the methoxyflurane Inhaler, with or without the AC chamber, creates additional risk. Elevation of liver enzymes, blood urea nitrogen, and serum uric acid, have been reported in healthcare professionals regularly exposed to methoxyflurane inhalational products. 8 A formal limit regarding levels of occupational exposure to methoxyflurane has not been established.

The risk of occupational exposure of methoxyflurane will be evaluated in a controlled laboratory setting, recruiting 30 health, screened (history and blood work) volunteers to participate in the back of an ambulance which meets the Ontario Ministry of Health Standards. The participants will consent and follow a protocol while active samplers are placed in the rear of the ambulance to capture the off-gassing of the methoxyflurane. This will inform the risk of occupational exposure of methoxyflurane to paramedics, as well as, hoping to inform the risk of multiple administrations by paramedics to different patients during a single shift, to ensure a medical directive can be created to support patient care and evaluate and support paramedic safety.

DETAILED DESCRIPTION:
Background:

Pain is a common emergency that is responsible for approximately 40% of ambulance calls.1 Effective and safe relief of acute pain is not only an important medical problem; since 2004, it is has been considered a fundamental human right.2 Yet, it is often undertreated in both prehospital and emergency department (ED) settings.3,4 Unrelieved pain activates the pituitary-adrenal axis, which can suppress the immune system and result in infection and poor wound healing. 5 Sympathetic activation can have negative effects on the cardiovascular, gastrointestinal, and renal systems, predisposing patients to adverse events such as cardiac ischemia.5 In addition, inadequate pain management is associated with physiological and psychological stress, which can impact therapy and rehabilitation, resulting in diminished quality of life of the patient.6 Drugs such as nonsteroidal anti-inflammatory drugs, ketamine, nitrous oxide, and opiates are widely used to manage acute pain by paramedics.7 Many of these treatments require higher level of paramedic training to administer, and require expensive equipment, peripheral intravenous access and titration of analgesia, which can be difficult without eliciting side effects.

Methoxyflurane belongs to the fluorinated hydrocarbon group of volatile anesthetic gases and was recently approved in Canada for emergency relief of pain associated with trauma in conscious adult patients. Methoxyflurane has analgesia properties at low doses and is rapidly absorbed into the bloodstream to produce analgesia.14 This inhalational analgesic has been used extensively in emergency settings in Australia and New Zealand for over 30 years. 13 Low-dose methoxyflurane is self-administered by patients in analgesic doses, at a maximum of two 3 mL doses of methoxyflurane 99.9%, in a single administration via a handheld inhaler (a green, whistle-shaped, single-use device).8-11 Methoxyflurane is added to the inhaler via a one-way valve and is absorbed by a polypropylene wick. Following instruction from a trained health care provider, the patient inhales the vaporized liquid through the mouthpiece and exhales back into the mouthpiece. Exhaled methoxyflurane is captured by an activated carbon (AC) chamber fitted to the inhaler in order to minimize environmental and occupational exposure. If stronger analgesia is required, the patient can cover the dilutor hole on the AC chamber. In vitro testing indicates that methoxyflurane concentrations delivered by the Penthrox® inhaler can reach a peak of 0.7% when the dilutor hole on the AC chamber is closed, and methoxyflurane concentrations are reduced by approximately 20% when the dilutor hole is open. 12 It provides rapid (<1 minute), short-term (30-45 minutes) pain relief within six to ten inhalations8 and has been shown to be effective and safe in emergency care13-16 and for minor surgical, radiological, and dental procedures.9,17

Methoxyflurane was first introduced to clinical practice as an inhalation anaesthetic in 1960. 18 Its clinical use as an anaesthetic was discouraged in the late 1970s to early 1980s due to the availability of newer anaesthetic agents and reports of dose-related renal tubular damage following prolonged exposure to this fluorinated hydrocarbon, thought to be caused by elevated levels of inorganic fluoride. 7,8,19 This led to its reduced use and disappearance from anaesthetic practice by the late 1970s before being voluntarily withdrawn from the markets in the Canada and the United States in the 1990s. 7-9 However, methoxyflurane was never withdrawn in Australia and New Zealand where it has been available as Penthrox® for use in lower doses as a rapid-acting analgesic for short-term pain relief. The lower analgesic doses of methoxyflurane in laboratory and clinical data indicated no increased risk of renal tubular damage.8 Since 1975, over five million methoxyflurane doses have been supplied. It is used by ambulance services, first responders as a first-line analgesic agent and in brief surgical procedures such as colonoscopies, bone marrow biopsies and changing of wound dressings. From laboratory studies and some clinical data, lower analgesic doses of methoxyflurane, indicated no increased risk of renal tubular damage.20

Exposure to inhaled anaesthetics is commonly assessed using the minimum alveolar concentration (MAC). This is the concentration of inhaled anesthetic within the alveoli at which 50% of people do not move in response to a surgical stimulus. At ≤2 MAC-hours, methoxyflurane results in serum fluoride concentration ≤40 μmol/L which is not associated with renal toxicity.20 The current dosing recommendation is 3 ml bottle is vaporized into the methoxyflurane inhaler and on finishing the 3 ml dose, another 3 ml may be used, if needed. However, the frequency at which methoxyflurane treatment can be safely used by paramedics is not established. From the product monograph, a patient's maximum daily dose of 6 mLs and weekly 15 mLs of methoxyflurane. 8 The treatment course of methoxyflurane for patients should not be repeated at an interval of less than 3 months. 8 Low-dose methoxyflurane analgesic levels, in accordance with current treatment recommendations, results in methoxyflurane exposure of 0.6 MAC-hours, providing a 2.7 to 8-fold renal safety margin for renal toxicity. Despite the activated carbon chamber to capture the exhaled methoxyflurane, when paramedics are supervising patients receiving inhaled analgesia within a confined area (like the back of an ambulance), it is possible that a paramedic may experience intermittent exposure to methoxyflurane vapour. Multiple use of the methoxyflurane Inhaler, with or without the AC chamber, creates additional risk. Elevation of liver enzymes, blood urea nitrogen, and serum uric acid, have been reported in healthcare professionals regularly exposed to methoxyflurane inhalational products. 8 A formal limit regarding levels of occupational exposure to methoxyflurane has not been established. However, a maximum 8-hour time weighted average (TWA) exposure level of 15 ppm was derived based on extrapolation of nephrotoxicity data from anaesthetized patients receiving high-dose methoxyflurane.12 This benchmark is well above the methoxyflurane odour threshold of 0.13-0.19 ppm.12 While low levels of methoxyflurane exposure have been documented by hospital staff supervising patients using Penthrox® inhalers during painful procedures, 12,21 studies are lacking to inform occupational exposure of paramedics to methoxyflurane vapour during transport in the small, enclosed space of an ambulance.

The study team conducted a feasibility study before deciding to embark on this laboratory study and a larger-scale clinical evaluation. During the feasibility study, occupational exposure was assessed in a real setting with consented paramedics. As this study was conducted pragmatically during ambulance calls, study was unable to determine when methoxyflurane was going to be used. Therefore, despite 30 samples being placed in ambulances, our study analyzed seven samples. Two were field blanks (i.e. no methoxyflurane was used during the paramedic shift) and two samples were controls and were never open but went through analysis. For the remaining three samples, the time of administration was 20 minutes, 16 minutes and 10 minutes. Each sampler was evaluated on a 720 minute exposure period resulting in a mean concentration of 0.0912 ppm (minimum=0.0147 and maximum 0.186 ppm). No exposures above the maximum exposure limit (MEL) of 15 ppm (8 TWA) were noted. The field blanks as well as the controls recorded <3ng when analyzed. These findings are consistent with other studies12 which showed levels of vapour capture below the ceiling limit of 2 ppm. Frangos et al. reported a mean 8-hour TWA methoxyflurane exposure by flight paramedics to be 0.23 ppm without the activated charcoal chamber within a confined ambulance and well below the MEL of 15 ppm. 12 This real-world study, conducted in the prehospital setting in the back of an ambulance, showed well below safe levels of methoxyflurane vapour exposure to paramedics. However, there is still a gap in knowledge on understanding this exposure and the cumulative risk of methoxyflurane administered multiple times during a paramedic's shift.

II- OBJECTIVES The risk of occupational exposure of methoxyflurane will be evaluated in a controlled laboratory setting, using an ambulance which meets the Ontario Ministry of Health Standards. 22 This will inform the risk of occupational exposure of methoxyflurane to paramedics, as well as, hoping to inform the risk of multiple administrations by paramedics to different patients during a single shift, to ensure a medical directive can be created to support patient care and evaluate and support paramedic safety.

The aim of this non-clinical laboratory-controlled study is to evaluate the risk, considering a maximum exposure limit (MEL) of 15 ppm (8-hour TWA), of occupational exposure of methoxyflurane in the back of an enclosed ambulance with single and multiple events.

III- METHODS Design This is a phase other, Health Canada regulated, non-clinical occupational exposure laboratory study, where healthy human participants will inhale methoxyflurane and during which occupational exposure of methoxyflurane will be measured via strategically positioned samplers (active and passive) according to a pre-set protocol, including single and multiple consecutive events.

Setting The study will be conducted in the back of a ministry approved ambulance where, according to the Ontario Provincial Land Ambulance & Emergency Response Standard, (REF) it requires the ventilation system(s) be capable of providing a complete change of ambient air within the vehicle every 2.5 minutes with the vehicle static. Ventilation shall be separately controlled within each compartment.22 The approximate cubic meter volume in the driver and patient compartment is 15 m3. The front and rear compartment are separated by a bulkhead with a communication window between the driver compartment and patient compartment.

Participants Recruitment A plain (lay) language posting in English will be developed, using a template from the Ottawa Hospital Research Institute (OHRI). The Ottawa Hospital (TOH) corporate social media and work with OHRI's media leads to assist with posters and other TOH available advertising to recruit interested participants to the study. These digital postings will have a phone number and email for interested participants to contact the research team. A research team member will contact the interested participant and complete the primary screening process and consent the participant to participate in the study. A standard clinical trial informed consent form from OHRI will be used. Once consent is complete the research team will send the participant a link to a participant enrollment form, developed using Microsoft Forms, to complete. All information regarding study participants will be kept on a secure server on the TOH SharePoint for a minimum of 15 years, only accessible by the research study team members. If the participant meets the primary screening criteria, has consented and has completed the enrollment form, they will move onto the secondary (laboratory) screening process.

Screening A standard protocol for screening the participants will be used. See flow diagram (appendix 1) for details. Inspiratory capacity and expiratory reserve volumes are similar among males ages ≥18 similarly among females ≥18.23 Therefore, age is not considered to bias or impact study results. Equal distribution across sexes when enrolling volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age

Exclusion Criteria:

* previous history of significant liver disease (e.g. Cirrhosis) or lab values outside normal range *;
* cardiac or respiratory illnesses (e.g. ischemic heart disease, asthma, chronic obstructive pulmonary disease/smoking hx >10 pack per year history);
* any renal impairment or lab values outside normal *;
* previous possible allergy to methoxyflurane by the patient or a
* drug interactions: concurrent use of any potential nephrotoxic drugs relative; (aminoglycosidese.g. gentamicin), colistin, polymyxin B, amphotericin B, and tetracyclines);
* personal or family history of malignant hyperthermia;
* inclusion in another study not allowing the co-enrollment;
* pregnancy or breastfeeding;
* and history of use of methoxyflurane in the last 3 months.

  * normal laboratory values will be determined based on The Ottawa Hospital's available reference ranges.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
8 hour Time weighted average | 15 minutes
  Eight-hour time weighted average (TWA) for methoxyflurane exposure level following a single participant protocol (1 event)
8 hour time weighted average | 120 minutes
  Eight-hour TWA for methoxyflurane exposure resulting from multiple participant protocols (multiple events)

SECONDARY OUTCOMES:
8 hour time weighted average | 15 minutes
  Eight-hour TWA for methoxyflurane exposure level following a single administration (ventilation off)
8 hour time weighted average | 15 minutes
  Eight-hour TWA for methoxyflurane exposure resulting from multiple participant protocols (ventilation off)
adverse events | 60 minutes
  Adverse events post administration of methoxyflurane: any advanced airway interventions, oxygen requirement (oxygen saturations <94%), drop in blood pressure by 40% and/or <90 systolic requiring intervention, malignant hyperthermia reaction
vital signs for participants | 60 minutes (5 minute interval)
  Other respiratory measures will be captured using ETCO2
vital signs for participants | 60 minutes (5 minute interval)
  estimating tidal volumes
vital signs for participants | 60 minutes (5 minute interval)
  respiratory rate
vital signs for participants | 60 minutes (5 minute interval)
  Heart Rate
vital signs for participants | 60 minutes (5 minute interval)
  blood pressure
vital signs for participants | 60 minutes (5 minute interval)
  oxygen saturation
vital signs for participants | 60 minutes (5 minute interval)
  temperature
vital signs for participants | 60 minutes (5 minute interval)
  level of responsiveness (Glasgow Coma Scale)
Residual methoxyflurane in the inhaler | 15 minutes
  Residual methoxyflurane in the inhaler

OTHER OUTCOMES:
environmental factors | 15 minutes
  Monitor temperature inside the ambulance (evaluated with and without the ventilation system).
environmental factors | 15 minutes
  Humidity inside the ambulance (evaluated with and without the ventilation system).

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Michael A Austin, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The health volunteers data is not part of the primary study, data regarding the volunteers will be aggregate and published in journals for other researches to review if appropriate.